CLINICAL TRIAL: NCT00081835
Title: Evaluation and Treatment of Ocular Complications of Vaccinia Vaccination: Suitability of NP-016 Vaccinia Immune Globulin (VIG) for Sight-Threatening Conditions [VIG31]
Brief Title: Evaluation and Treatment of Eye Complications of Vaccinia Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040157; 04-EI-0157
Record Dates: First submitted 2004-04-22; First posted 2004-04-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-08-15

CONDITIONS: Vaccinia
Keywords: Smallpox; Cowpox; Corneal Ulcer; Keratitis; Immune Response, Vaccine; Cornea; Vaccinia; Vaccinia Immune Globulin (VIG); Conjunctivitis; Vaccinia Vaccination; Smallpox Vaccination
MeSH Terms: conditions — Vaccinia; Smallpox; Cowpox; Corneal Ulcer; Keratitis; Corneal Diseases; Conjunctivitis

INTERVENTIONS:
Drug: NP-016 Vaccine Immune Globulin (IV-VIG)

SUMMARY:
This study will evaluate patients with eye complications related to vaccination against smallpox to learn more about these conditions. Vaccinia vaccination has been used for more than 100 years for preventing smallpox. A small number of people who receive the vaccination (less than 1 in 1,000) develop complications, sometimes in their eyes. This usually results from the accidental transfer of the infection from the vaccination site to the face or eyes, perhaps by touching the vaccination area and then the face or eyelids before washing the hands. The study will also examine whether an experimental treatment called NP-016 vaccinia immune globulin can reduce corneal scarring that is sometimes associated with serious vaccinia complications and can impair vision.

Children and adults with keratitis, severe conjunctivitis, or blepharitis following exposure to vaccinia vaccination may be eligible for this study. Children must weigh at least 10 kg.

Participants undergo the following tests and procedures at enrollment, with some tests repeated at scheduled study visits:

1. Medical history and physical examination
2. Infectious disease consultation
3. Complete eye evaluation including:

   * Fundus photography to examine the back of the eye - dilation of the pupils with eye drops to examine and photograph the back of the eye
   * Slit lamp biomicroscopy - evaluation of the front part of the eye with a slit lamp microscope
   * Eye pressure measurements
   * Eye swab to look for vaccinia virus or other causes of disease
4. Blood tests
5. Photographs and documentation of eye and skin lesions
6. Vaccinia diagnostic tests, such as skin or mucosa scrapings; blood, throat, or urine cultures; and tissue biopsies, if needed

Patients begin treatment with standard medications for their eye disease, such as trifluridine (Viroptic® (Registered Trademark)) anti-viral eye drops. Patients whose condition becomes serious are offered additional treatment with intravenous (through a vein) infusions of either VIG or placebo (salt water solution with no active drug) and are randomly assigned to one or the other treatment group. All patients continue standard-of-care treatment as well.

Follow-up visits at the NIH eye clinic are scheduled as required by the patient's condition. Patients with mild complications who are taking only standard medications may need to be seen only 1 month after the initial visit and then 6 months and 12 months later. Patients with more serious conditions who qualify for VIG or placebo treatments may be seen daily for a week, then once a week for the rest of the first month, and then at 6 months and 12 months, unless more frequent treatment or observation is required.

DETAILED DESCRIPTION:
Vaccinia virus (a live but relatively weak relative of smallpox and cowpox) is used to vaccinate people against the development of smallpox (variola) resulting from an infection with the viral genus Orthopoxvirus. Although, smallpox was thought to be eradicated worldwide during the 1970's, some smallpox cultures have been retained in the laboratories of several countries and may pose a potential threat if used as a biological weapon. This has recently led to programs where mass-inoculations with vaccinia have been initiated throughout the U.S.

Vaccination against smallpox using vaccinia can result in complications. Reactions are rarely serious or life threatening, but one of the most common serious complications occur in and around the eye. This occurs when a person transfers vaccinia viruses by touch from their primary inoculation site to their own eyes (auto-inoculation). Accidental exposure can also occur in the laboratory or by contact with a vaccinated person. Ocular involvement may be confined to the lids or conjunctiva but may easily be transferred to the cornea. Keratitis can result in scarring that could have a severe and permanent impact on vision. Even when the cornea is not affected, extensive lesions on the lid or other ocular tissues can lead to additional sight-threatening complications.

Recently, the US Food and Drug Administration licenced Vaccinia Immune Globulin Intravenous (Human) (VIGIV, formerly known as NP-016). It is indicated for the "treatment and/or modification of the following conditions, which are complications resulting from smallpox vaccination: (a) Eczema vaccinatum; (b) Progressive vaccinia; (c) Severe generalized vaccinia; (d) Vaccinia infections in individuals who have skin conditions such as burns, impetigo, varicella-zoster, or poison ivy; or individuals who have eczematous skin lesions because of either the activity or extensiveness of such lesions; and (e) Aberrant infections induced by vaccinia virus that includes its accidental implantation in eyes (except in cases of isolated keratitis), mouth, or other areas where vaccinia infection would constitute a special hazard." The precautionary statement regarding isolated vaccinia keratitis appears though it is uncertain whether VIGIV use will decrease or increase corneal scarring in humans. The implication of increased scarringis based on some evidence in animal models indicating that more extensive corneal clouding can occur following VIG therapy. To investigate if this implication has clinical significance, two hundred study participants with corneal involvement following vaccinia vaccination or other exposure will be randomized to receive either placebo or VIGIV. All enrolled participants will be provided standard-of-care antiviral treatments for ocular complications. One-year proportions of corneal scarring will be compared between the two groups. Further knowledge about the biologic mechanisms of complications associated with vaccinia vaccination and rapid diagnostic test may lead to more effective forms of therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to enroll in this study, a prospective participant must satisfy all of the following inclusion criteria:

1. The participant, or their parent or guardian if younger than 18 years at enrollment, is able to understand and sign an approved consent form. Any minor participant with adequate reading and writing skills must also sign an assent using a form approved by the local Institutional Review Board or Independent Ethics Committee (IRB/IEC). Minors with verbal skills but without adequate reading and writing skills should have an acknowledgement signed by their parent or guardian to certify that verbal assent to participate was obtained.
2. The participant must have received the vaccinia vaccination, been exposed to a person vaccinated with vaccinia who has skin lesions, or been exposed directly to accidental splash of the vaccine.
3. Have signs and symptoms consistent with ocular vaccinia.
4. To be eligible for randomization the participant must have corneal involvement defined as a keratitis with any abnormality of the epithelium, stroma, or endothelium consistent with vaccinia infection.

EXCLUSION CRITERIA:

To be randomized to the VIGIV/placebo treatment, a proposed participant must not satisfy the following exclusion criteria:

1. Children with body weight less than 10 kg.
2. Have a known severe reaction to the IV or IM administration of human immunoglobulin.
3. Have known severe acute allergic reactions to the non-active ingredients of polysorbate 80, maltose, or the trace amounts of TNBP or Triton X-100 used in the preparation of VIGIV.
4. Has received VIGIV within 6 months prior to randomization.
5. Pregnant women, unless an approved, specific additional consent statement attesting to awareness of the unknown risk of VIGIV therapy during pregnancy is understood and signed by the participant.
6. Have orbital cellulites.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2004-04-19; Study Completion 2007-08-15

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ruben FL, Lane JM. Ocular vaccinia. An epidemiologic analysis of 348 cases. Arch Ophthalmol. 1970 Jul;84(1):45-8. doi: 10.1001/archopht.1970.00990040047012. No abstract available. PMID 5423606